CLINICAL TRIAL: NCT02119611
Title: Deep Brain Stimulation Therapy in Movement Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140086; 14-N-0086
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-07

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation; Movement Disorders; Parkinson's Disease; Essential Tremor; Tourette Syndrome
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Essential Tremor; Tourette Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Other): Therapy
  Interventions: Device: Deep Brain Stimulation management

INTERVENTIONS:
Device: Deep Brain Stimulation management — The DBS surgery will be performed according to standard of care in the centers of referral. If performed at the NIH, this will be done under protocol 11-N-0211 or other protocols permitting DBS surgery depending on future availability.

SUMMARY:
Background:

- In deep brain stimulation (DBS), a device called a neurostimulator is placed in the chest. It is attached to wires in parts of the brain that affect movement. DBS might help people with movement disorders like Parkinson s disease (PD), dystonia, and essential tremor (ET).

Objective:

- To provide DBS treatment to people with some movement disorders.

Eligibility:

- Adults 18 years and older with PD, ET, or certain forms of dystonia.

Design:

* Participants will be screened with medical history and physical exam. They will have blood and urine tests and:
* MRI brain scan. The participant will lie on a table that slides in and out of a metal cylinder with a magnetic field. They will be in the scanner about 60 minutes. They will get earplugs for the loud noises. During part of the MRI, a needle will guide a thin plastic tube into an arm vein and a dye will be injected.
* Electrocardiogram. Metal disks or sticky pads will be placed on the chest, arms, and legs. They record heart activity.
* Chest X-ray.
* Tests of memory, attention, concentration, thinking, and movement.
* Eligible participants will have DBS surgery. The surgery and hospital care afterward are NOT part of this protocol.
* Study doctors will see participants 3 4 weeks after surgery to turn on the neurostimulator.
* Participants will return every month for 3 months, then every 3 months during the first year, and every 6 months during the second year. Each time, participants will be examined and answer questions. DBS placement will be evaluated with MRI. The neurostimulator will be programmed. At two visits, participants will have tests of movements, thinking, and memory.

DETAILED DESCRIPTION:
Objective

The purposes of this protocol are:

To provide DBS therapy and follow-up management

To maintain a cohort of patients treated with DBS who can participate in other NIH protocols addressing the efficacy of functional surgery and the relevant physiology.

To collect physiology, programming, and efficacy data related to DBS therapy and motor and cognitive function in these patient populations. All the data collected will be an outcome of standard of care and all analyses will be retrospective.

All treatment under this protocol will be based on the current standard of care for DBS therapy. All tests and study procedures will be administered per standard and routine clinical care; however, the schedule of procedures has been standardized for research purposes. Subjects may be enrolled in the study to support participation in other DBS protocols.

Study Population

Patients 18 years and older with medically refractory PD, dystonia, and/or ET may participate in this study. Other indications will be added with subsequent amendments if FDA approval of deep brain stimulation is extended to other conditions.

Study Design

The treatment that is rendered in this protocol is standard of care for PD, dystonia, and ET. Patients confirmed to have medically refractory PD, dystonia or ET will be offered DBS as a therapeutic option per standard of care procedures and routine clinical care. Patients will be evaluated for their eligibility for the procedure and the risk/benefit balance for surgical therapy will be assessed (Lang et al., 2006). After completing the evaluation, a decision will be made on recommending the procedure. At that point the patients will be referred for the surgical intervention to the NIH Surgical Neurology Branch or to collaborating surgeons in the community. If the surgery is performed at the NIH, the Neurology DBS team can be involved in surgical planning, target selection, intraoperative physiology recording and testing, as specified under SNB protocols. After the surgery, the patients will be followed in the NIH DBS clinic and the DBS programming will be initiated and performed as outlined below. The patients will be followed up for at least two years, and then they will have the option to transfer their care back to the neurologists in the community or continue care with the NIH Neurology team until care in the community is available.

In addition, patients can be enrolled in the protocol at various points in relation to DBS surgery.

Data regarding the movement disorder of the subject and observations of their standard of care treatment will be collected. Data may be used for future research questions that are related to subjects movement disorder and/or treatment.

Outcome Measures

1. To evaluate effects of DBS before and after surgery using clinically-generated data on:

   1. Severity of PD motor symptoms (measured by the UPDRS III scale)
   2. Changes in dystonia severity (measured by the Burke-Fahn-Marsden (BFM) dystonia rating scale (Burke et al., 1985)
   3. Changes in tremor severity (measured by the Tremor Rating Scale (TRS))
   4. Levels of effective drug therapy for PD patients using the Levodopa Equivalent Drug Dosing (LEDD)
   5. Changes in behavior, performance of activities of daily living and complications of therapy as measured by the UPDRS I, II, and IV scales
2. To evaluate effects of DBS before and after surgery on quality of life:

   1. For PD patients (measured by UPDRS part II and other scales such as the PDQ-39)
   2. For the Dystonia and ET patients (measured by the SF-12 scale)
3. To evaluate radiographic correlation of DBS electrode position and clinical changes
4. To evaluate neurophysiological mechanisms of DBS and relevant basal ganglia physiology

All data collected will be done as standard of care and all analysis will be retrospective.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, candidates must meet all the following criteria:

* Be 18 years of age or older.
* Able to comply with study procedures and provide informed consent.
* Have a clinical diagnosis of idiopathic PD, primary dystonia, or ET:

  1. The diagnosis of idiopathic PD will be based on the UK Brain Bank Criteria, and confirmed by the Movement Disorders Neurologists in the NIH Parkinson Clinic.
  2. The diagnosis of primary (generalized or segmental), hemidystonia, or cervical dystonia will be confirmed on clinical examination in the NIH Movement Disorders Clinic.
  3. The diagnosis of ET will be confirmed on clinical examination in the NIH Movement Disorders Clinic (the diagnosis of ET will be based on bilateral, largely symmetric postural or kinetic tremor involving hands and forearms that is visible and persistent. Additional or isolated tremor in head may be present but there should be the absence of abnormal posturing).
* a. History of appropriate response to dopaminergic medication, with at least a 30% improvement in motor UPDRS with L-DOPA by history or in-clinic testing, for the PD patients. OR

  b.Patients with tremor-dominant PD that do not respond to dopaminergic therapy and that exhibit a tremor score of at least 2 for tremor severity on at least one side of the body on the motor UPDRS examination.
* Unsatisfactory clinical response to maximal medical management (with trials of both higher and lower doses of drugs), including:

For PD patients:

1. good benefit from dopaminergic medication but associated with insufficient duration of action or unacceptable side-effects OR
2. intractable disabling motor fluctuations (severe off periods, dyskinesias, or freezing spells) OR

   For ET and dystonia:
3. intractable symptoms of ET or dystonia impacting at least 2 activities of daily living.

   * Interested in being evaluated to undergo DBS, if indicated, to treat medically refractory movement disorder or
   * Patients already implanted with DBS for continued management

(Note: Inclusion criteria 4 and 5 can be met by historical report in patients who had DBS implanted outside the NIH)

EXCLUSION CRITERIA:

For those who have not had DBS:

Candidates will be excluded if they meet any of the following criteria:

* Clinically significant medical disease that would increase the risk of developing pre- or postoperative complications, including but not limited to uncontrolled systemic hypertension with values above 170/100; unstable heart disease; unstable respiratory disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation which cannot be interrupted;
* Evidence of secondary or atypical parkinsonism/dystonia/tremor as suggested by:

  1. History of stroke, exposure to toxins, neuroleptics, or encephalitis
  2. Neurologic signs of upper motor neuron or cerebellar involvement, supranuclear gaze palsy, or multiple systems atrophy.
  3. MR-imaging with evidence indicative of secondary disease such as tumor, or stroke, which could cause the movement disorder.
* Dementia as evidenced by formal neuropsychological evaluation, Mattis Dementia Rating Scale (DRS-2) score, and clinical evaluations.
* Unable to complete cognitive assessments and testing necessary to adequately evaluate risks and benefits of surgery.
* Clinically signficiant or unstable psychiatric disorder such as severe depression or anxiety, which, in the opinion of the investigators would increase the risk of developing postoperative complications.
* Unable to undergo MR-imaging because of implanted pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal workers may have, or if candidates are uncomfortable in small closed spaces (have claustrophobia), or cannot lie comfortably on their back for up to one hour.
* Pregnant women.
* Otherwise not eligible for DBS surgery, for example known inability to undergo anesthesia

For those who have had DBS:

-Contra-indications for ongoing stimulation, such as intractable side effects of DBS despite stimulation parameter adjustment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-04-02 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
To provide DBS therapy and follow-up management | two years
  a. Severity of PD motor symptoms (measured by the UPDRS III scale) b. Changes in dystonia severity (measured by the Burke-Fahn-Marsden (BFM) dystonia rating scale (Burke et al., 1985) c. Changes in tremor severity (measured by the Tremor Rating Scale (TRS)) d. Levels of effective drug therapy for PD patients using the Levodopa Equivalent Drug Dosing (LEDD) e. Changes in behavior, performance of activities of daily living and complications of therapy as measured by the UPDRS I, II, and IV scales 2. To evaluate effects of DBS before and 1 year after surgery on quality of life: a. For PD patients (measured by UPDRS part II and other scales such as the PDQ-39) b. For the Dystonia and ET patients (measured by the SF-12 scale) 3. To evaluate radiographic correlation of DBS electrode position and clinical changes 4. To evaluate neurophysiological mechanisms of DBS and relevant basal ganglia physiology
To maintain a cohort of patients treated with DBS who can participate in other NIH protocols addressing the efficacy of functional surgery and the relevant physiology | ongoing
  To potentially enroll subjects in other NIH studies.
Data collection | ongoing
  All the data collected will be an outcome of standard of care and all analyses will be retrospective

SECONDARY OUTCOMES:
To access other clinical outcome measures related to response to therapy | 2 years
  Data collection
To correlate radiographic data related to DBS electrode position with clinical changes | 2 years
  Data collection
To collect physiology data correlated with motor and cognitive function in these | 2 years
  Data collection

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The DBS programing and management provided in this protocol is standard of care and all data is obtained in the course of standard of care treatment and data will be analyzed retrospectively. Since many patients continue to receive ongoing care through this protocol, it is unclear whether it will be feasible to make individual patient data available. This will likely depend on the specific analysis and result.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-N-0086.html